CLINICAL TRIAL: NCT00556569
Title: Evaluation of CHAM JAM (Previously Known as the Moving Smart) Intervention in Increasing Physical Activity in Bronx Elementary School Students
Brief Title: Evaluation of CHAM JAM Increasing Physical Activity Levels in Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Philip O. Ozuah, Principal Investigator, Montefiore Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 07-08-253; RC1HD063607 (NIH)
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Physical Activity; Obesity
Keywords: Physical activity; Obesity
MeSH Terms: conditions — Motor Activity; Obesity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): 2 Intervention schools are cluster randomized to receive CHAM JAM (previously known as the Moving Smart Program) in Year 1
  Interventions: Other: CHAM JAM
- Wait-Listed Control (No Intervention): 2 Wait-Listed Control Schools will receive CHAM JAM (previously known as the Moving Smart Program) in Year 2 of the study

INTERVENTIONS:
Other: CHAM JAM — CHAM JAM (previously known as Moving Smart" (MS) program) is a daily, 10-minute classroom-based physical activity program led by teachers that integrates academic objectives with physical activity
  Other Names: Moving Smart Program; exercise program
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine if the "Moving Smart" program, a daily 10-minute classroom-based exercise program, increases physical activity levels during the school day in Bronx elementary school students.

DETAILED DESCRIPTION:
Background: Medical and national public health authorities recommend daily school physical education for all ages due to well-known health benefits of physical activity. Nevertheless, daily physical education among elementary and secondary school students is not common in United States' (US) schools. Moreover, some of the schools in many US cities, such as the Bronx, do not even have gymnasiums or physical education teachers.

Objective: We propose to implement and test the effectiveness and feasibility of the "Moving Smart" (MS) program, a daily, 10-minute classroom-based physical activity program led by teachers that integrate academic objectives with physical activity, on increasing physical activity (PA) levels during the school day in Bronx elementary school students.

Design/ Methods: A cluster-randomized, wait-listed control trial of four Bronx elementary schools with one-year follow-up longitudinal study. Students in two intervention schools will receive the MS 3-times daily, for 10-minutes each time, in addition to regular physical education classes. Two wait-listed control schools will receive their regular physical education classes only. Subjects in the wait-listed control group will be offered the MS after the program is withdrawn from the intervention group at the end of the first year of study. A pedometer, an objective measure of PA in children, will be used to determine mean number of steps each student takes during school hours for 5 consecutive days at baseline, and every 3-months during the 2-year study period. For longitudinal follow-up, we will collect data from intervention group students and teachers on PA levels every 3-months for one-year after the intervention cessation. We will also collect yearly BMIs as a measure of overweight status. Descriptive statistics will be used to portray baseline characteristics of each group based on school, district, region, and NYC-wide data. The impact of the intervention on PA will be measured by comparing intervention and control schools using pedometer measurements as the primary dependent variable and students as the unit of analysis. We will collect fidelity measures by randomly selecting classes from the intervention schools and directly observing the level of PA present. We will determine the extent to which the MS becomes a part of the routine school policy by following the students and teachers from the intervention schools for 1-year after the intervention cessation.

ELIGIBILITY:
Inclusion Criteria:

* Elementary school students in K-3 grade in the Bronx, New York

Exclusion Criteria:

* Inability to participate in basic exercise program
* Students whose parents signed the opt-out letter

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10098 (Actual)
Dates: Start 2007-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
pedometer-derived step count | baseline and every 3 months
  mean number of step counts

SECONDARY OUTCOMES:
Body mass index | baseline and 1 year later
  formula for BMI that includes weight and height

OTHER OUTCOMES:
Fitness assessment for subset of students | baseline, 3 months and 12 months
  FitnessGRAM and step test

CONTACTS AND LOCATIONS:
Overall Officials: Philip O Ozuah, M.D., Ph.D., Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- 4 Elementary Schools, The Bronx, New York, United States

REFERENCES:
- [Result] Reznik M, Wylie-Rosett J, Kim M, Ozuah PO. A classroom-based physical activity intervention for urban kindergarten and first-grade students: a feasibility study. Child Obes. 2015 Jun;11(3):314-24. doi: 10.1089/chi.2014.0090. Epub 2015 Mar 6. PMID 25747719
- [Result] Reznik M, Wylie-Rosett J, Kim M, Ozuah PO. Physical activity during school in urban minority kindergarten and first-grade students. Pediatrics. 2013 Jan;131(1):e81-7. doi: 10.1542/peds.2012-1685. Epub 2012 Dec 3. PMID 23209101